CLINICAL TRIAL: NCT05423925
Title: Comparison of Perioperative Outcome Between Monopolar and Bipolar Hysteroscopic Myomectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 111121-E
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Hysteroscopic Myomectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- monopolar: monopolar electrodes, and have their corresponding distension media.
  Interventions: Procedure: Monopolar hysteroscopic myomectomy
- bipolar: bipolar electrodes, and have their corresponding distension media.
  Interventions: Procedure: Bipolar hysteroscopic myomectomy

INTERVENTIONS:
Procedure: Bipolar hysteroscopic myomectomy — Bipolar hysteroscopic myomectomy.
  Groups: bipolar
Procedure: Monopolar hysteroscopic myomectomy — Monopolar hysteroscopic myomectomy
  Groups: monopolar

SUMMARY:
Objective:

To evaluate clinical outcome between monopolar and bipolar hysteroscopic myomectomy.

DETAILED DESCRIPTION:
Methods:

Hysteoscopic myomectomy is a safe and effective procedure to remove submucosal myoma. Distension media is needed to distend the uterine cavity during the procedure. The electric cutting loops included monopolar and bipolar electrodes, and have their corresponding distension media. Medical records, including outpatient and inpatient records, operation note, and laboratory data, of all consecutive women who received hysteroscopic myomectomy between July 2008 and April 2022 will be reviewed.

Expected result: The investigatorscan get the differences between monopolar and bipolar hysteroscopic myomectomy, and the result can be used as a reference in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* women who received hysteroscopic myomectomy between July 2008 and April 2022 will be reviewed.

Exclusion Criteria:

* < 20 years old women
* Cervical fibroids were excluded.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women who received hysteroscopic myomectomy between July 2008 and April 2022 will be reviewed.
Study Population: > 20 years old women who received hysteroscopic myomectomy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Infused volume of distension medium | 3 months
  The differences of infused volume of distension medium

SECONDARY OUTCOMES:
Operation time | 3 months
  The between-group difference in operation time
Pain score after the procedure | 3 months
  The between-group difference in pain score after the procedure Pain score:0-10, the minimun values mean a better

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No